CLINICAL TRIAL: NCT06467851
Title: An Interventional Clinical Study to Investigate the Effect of Oral Administration of Suanzaoren Decoction and Huanglian Wendan Decoction on Human Biorhythms in Patients With Insomnia
Brief Title: Effect of Suanzaoren Decoction and Huanglian Wendan Decoction on Biorhythm of Insomnia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-431
Record Dates: First submitted 2024-06-16; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Chronic Insomnia; Melatonin; Circadian Rhythm; Suanzaoren Decoction and Huanglian Wendan
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subject group (No Intervention): Healthy subjects completed questionnaires and underwent saliva collection
- Chronic insomnia patients group (Experimental): Questionnaire completion and saliva collection in patients with chronic insomnia before and after Chinese herbal medicine treatment, respectively
  Interventions: Drug: Suanzaoren Decoction and Huanglian Wenda Decoction

INTERVENTIONS:
Drug: Suanzaoren Decoction and Huanglian Wenda Decoction — Twice daily. Chinese herbal medicine includes: 25 grams of Suanzaoren, 10 grams of chuanxiong, 30 grams of fushen, 10 grams of Polygala tenuifolia, 10 grams of Pinellia ternata, 12 grams of tangerine peel, 15 grams of Zhuru, 30 grams of forged keel, 30 grams of forged oyster,10 grams of aurantii fructus, 6 grams of coptis chinensis, 30 grams of Albizzia bark.Add or subtract Chinese herbal medicine according to the different clinical manifestations of each patient.
  Arms: Chronic insomnia patients group

SUMMARY:
The purpose of this study was to examine the impact of Chinese medicine on melatonin levels in patients with insomnia

DETAILED DESCRIPTION:
This was a single-centre, non-randomised, interventional study with a planned enrolment of 20 subjects, including 10 Chinese insomnia patients and 10 healthy subjects. All subjects giving written informed consent. Healthy subjects were admitted to the study ward at baseline (D-3), completed the Pittsburgh Sleep Quality Index (PSQI), Morning and Evening Questionnaire (MEQ), and began saliva collection at 16:00, stayed overnight in the study ward that night and were discharged the following day (D-2). Insomnia patients were admitted to the study ward at baseline (D-3), completed the PSQI and MEQ questionnaires and started saliva collection at 16:00, stayed overnight in the study ward and left the following day (D-2) after completing the relevant examinations. After 4 weeks of treatment with Suanzaoren Decoction and Huanglian Wendan Decoction, the subject was re-admitted to the study ward on D30, completed the PSQI and MEQ questionnaires and started saliva collection at 16:00, stayed overnight in the study ward and left on the following day (D31) after completing the relevant examinations. The intervention for patients with insomnia in this study was the administration of Suanzaoren Decoction and Huanglian Wendan Decoction twice a day for 4 weeks. Add or subtract Chinese herbal medicine according to the different clinical manifestations of each patient.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55, male or female；
* Insomnia patients: patients who met the diagnostic criteria for insomnia in the Chinese Guidelines for the Diagnosis and Treatment of Insomnia in Adults (2017 edition) and who were judged to have moderate-to-severe insomnia according to the Insomnia Severity Index Scale; Healthy subjects: those who had normal sleep, and who met the scores of 0 to 7 on the Insomnia Severity Index Scale;
* Informed consent, voluntary participation in the study；

Exclusion Criteria:

* People with mental illness;
* Chronic insomnia with yang deficiency and yin deficiency, clinical manifestations: coldness of the whole body and hands and feet, like warmth and pressing, yellowish colour, unshaped stools, lumbago, weakness of the legs, nocturia, pale tongue with thin white moss;
* Pregnant, lactating women;
* Have a serious primary heart, liver, lung, kidney, haematological or serious disease affecting their survival, e.g. tumour or AIDS, SCr > 1.5N (N is the upper limit of normal), ALT > 2N (N is the upper limit of normal), blood leucocytes < 3.0 x 109/L;
* Participants in any other clinical trial within 3 months prior to dosing;
* Those who are vulnerable to missing visits based on other circumstances that the researcher judges to be unsuitable for enrolment, such as changes in the work environment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in melatonin concentration at Week 4 | Baseline and Week 4
  The level of melatonin in the body

SECONDARY OUTCOMES:
Change from Baseline in the total score of the Pittsburgh sleep quality index (PSQI) at 4 weeks | Baseline and Week 4
  The Pittsburgh sleep quality index (PSQI) is a validated,self-reported instrument assessing the sleep quality over the past 4 week period. Possible scores range from 0(the best sleep quality) to 21(the worst possible sleep) quality).The higher the score of PSQI, the worse the sleep quality. Change=(Month 1 Score-Baseline Score)
Change from Baseline in the total score of Morning and Evening Questionnaire (MEQ) at 4 weeks | Baseline and Week 4
  The Morning and Evening Questionnaire (MEQ) was used to evaluate the type of biological clock of subjects

CONTACTS AND LOCATIONS:
Overall Officials: Xiuqin Wang, doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Feng Shao, doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No